CLINICAL TRIAL: NCT04994977
Title: Intra-Arterial (IA) Chemotherapy for Newly Diagnosed, Residual, or Recurrent Atypical Choroid Plexus Papilloma (ACPP) and Choroid Plexus Carcinoma (CPC) Prior to Second-Look Surgery
Brief Title: Intra-Arterial Chemotherapy for Newly Diagnosed, Residual, or Recurrent Atypical Choroid Plexus Papilloma and Choroid Plexus Carcinoma Prior to Second-Look Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-08022610
Record Dates: First submitted 2021-07-17; First posted 2021-08-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Atypical Choroid Plexus Papilloma; Choroid Plexus Carcinoma
MeSH Terms: conditions — Choroid Plexus Carcinoma | interventions — Melphalan; Carboplatin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intra-arterial Chemotherapy (Experimental): Subjects are pre-treated with heparin, and then given single doses of Melphalan, Carboplatin, and Topotecan consecutively via intra-arterial infusion. Multiple arteries may be used, with the total dose of the drugs remaining the same.
  Interventions: Drug: Melphalan; Drug: Carboplatin; Drug: Topotecan

INTERVENTIONS:
Drug: Melphalan — Given at 0.5 mg/ml.
Drug: Carboplatin — Given at 5 mg/ml.
Drug: Topotecan — Given at 0.2 mg/ml.

SUMMARY:
This study will test the safety and efficacy of intra-arterial chemotherapy in subjects with newly diagnosed, residual, or recurrent atypical choroid plexus papilloma and choroid plexus carcinoma prior to a second surgery.

It is believed that intra-arterial chemotherapy will be safe and feasible for this population and will result in decreased tumor size, which may further improve the goals of a second-look surgery.

DETAILED DESCRIPTION:
The intent of this study is to determine if intra-arterial chemotherapy is a safe and effective option for subjects with atypical choroid plexus papilloma and choroid plexus carcinoma prior to receiving second-look surgery. Angiography occurs when a catheter is inserted through the subjects vasculature to the major vessels that supply cerebral circulation. Subjects on this trial will undergo a a cerebral angiogram to determine the ideal arteries to use for drug infusion. Once identified, chemotherapy will be delivered through the catheter directly to the site of tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a histologically confirmed diagnosis of ACPP or CPC that is newly diagnosed, residual or recurrent.
2. Subjects must have a Karnofsky or Lansky Performance Score ≥ 60 % assessed within two weeks prior to enrollment. Karnofsky is used for patients ≥ 16 years and Lansky for those < 16.
3. Subjects must have normal organ and marrow function documented within 14 days of enrollment and within 7 days of the start of treatment as noted below:

   1. Absolute neutrophil count ≥ 1,000/μL
   2. Platelets ≥ 100,000/μL (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to enrollment)
   3. Hemoglobin ≥ 8 g/dL (may receive PRBC transfusions)
   4. Total bilirubin < 1.5 times upper limit of normal for age
   5. AST (SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal for age
   6. Creatinine clearance or radioisotope GFR ≥ 70 ml/min/1.73m2 or a serum creatinine WNL for age as determined using the Schwartz formula.36
   7. Sodium, Potassium, Calcium and Magnesium < 1.5x institutional ULN
   8. Albumin ≥ 3 g/dL
4. Subjects who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to enrollment.
5. Subjects with neurological deficits should have deficits that are stable for a minimum of 1 week prior to enrollment.
6. If the subject has any of the following therapies, must be at least:

   * 4 weeks post-focal RT (radiation therapy), 3 months post-CSI (craniospinal irradiation)
   * 4 weeks post-myelosuppressive chemotherapy (if post-nitrosoureas, must have 6 weeks therapy)
   * 4 weeks post-monoclonal antibodies
   * 1 week post-targeted therapy
7. If subject has received any previous treatment, all treatment related toxicities should have recovered to < grade 2
8. Subject or parent must sign a written informed consent document according to institutional guidelines.

Exclusion Criteria:

1. Females who are pregnant or lactating.
2. Subjects with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) likely to interfere with the study procedures or results.
3. Subjects who are receiving any other anticancer or investigational agents.
4. Subjects with uncontrolled seizures.
5. Subjects receiving enzyme inducing anticonvulsants.
6. Subjects with other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) including heart failure that meets New York Heart Association (NYHA) class II or above.
7. Subjects who have had an allogenic bone marrow transplant < 6 months prior to enrollment or an autologous bone marrow/stem cell transplant < 3 months prior to enrollment.
8. Subjects with multifocal disease or disease that has been disseminated will not be eligible for this study. They will undergo systemic chemotherapy and their disease will be further evaluated prior to be eligible for 2nd look surgery.
9. This study will only enroll subjects with ACPP or CPC and will not enroll subjects with choroid plexus papilloma (CPP). ACPP or CPC subjects with symptomatic hydrocephalus will not be eligible for this study. These subjects will have to be treated for their hydrocephalus and be re-evaluated according to our eligibility criteria in order to be enrolled.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety of intra-arterial chemotherapy in subjects with ACPP and CPC, measured by the number of serious adverse events that are reported as at least possible related to the intervention that occur in subjects on the trial | Through study completion, a little over a year for each subject

SECONDARY OUTCOMES:
The number of successful angiography procedures, determined by examination of vasculature and assessment of catheter placement | On Day 1 of the trial for each subject
The number of patients with a tumor volume reduction response, determined by MRI assessments | Between 4-6 weeks after intra-arterial chemotherapy
The proportion of patients with a tumor volume reduction response, determined by MRI assessments | Between 4-6 weeks after intra-arterial chemotherapy
The number of patients with a tumor vascularity reduction response, determined by MRI assessments | Between 4-6 weeks after intra-arterial chemotherapy
The proportion of patients with a tumor vascularity reduction response, determined by MRI assessments | Between 4-6 weeks after intra-arterial chemotherapy
The success of second look surgery determined by measuring the extent of tumor resection | Around 7 weeks after intra-arterial chemotherapy, during second look surgery
The success of second look surgery determined by amount of blood loss | Around 7 weeks after intra-arterial chemotherapy, during second look surgery
The success of second look surgery determined by percent of blood loss | Around 7 weeks after intra-arterial chemotherapy, during second look surgery

OTHER OUTCOMES:
Extent of pathology correlation to tumor vascularity and tumor viability | Around 7 weeks after intra-arterial chemotherapy
  Determined by comparison of pathology reports and surgical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Mark Souweidane, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No